CLINICAL TRIAL: NCT05328193
Title: Food for Thought: Virtual Home-Based Family Interventions to Improve Nutrition Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Joe C Davis Foundation (Unknown)
Responsible Party: Principal Investigator, Shari Barkin, MD, MSHS, Division Chief of Academic General Pediatrics, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 200257
Record Dates: First submitted 2022-03-30; First posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Behavior, Health; Obesity, Childhood
MeSH Terms: conditions — Health Behavior; Pediatric Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: All study personnel that are in a position to change the study protocol or its implementation in study participants should be blinded to information that may allow them to do so, from when the study starts until the study ends, with specific exceptions. This means that all investigators and study staff should be blinded to study data aggregated by study arm that have the potential to impact the study's outcome.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teaching Kitchen Outreach (Active Comparator): All participants (both the intervention and control condition) will receive to 11 weekly short (about 2-3 minutes) Teaching Kitchen Outreach (TKO) videos. Recipe specific groceries will be delivered to participants' homes by a third party grocery delivery company, or will be available for pickup at a central location(s). These recipes reflect foods that can be purchased with SNAP and WIC and include tested meals and snacks that were developed and evaluated in person in Parks and Recreation after-school programming.
  Interventions: Behavioral: Teaching Kitchen Outreach
- Healthier Families, COVID Edition (Experimental): Those randomized to the intervention condition will also receive a 12-weekly health coach via a virtual platform (such as Zoom, FaceTime, or What's App) to provide an adapted version of the previously tested Healthier Families program. Adaptations include: shortening each session to 30 minutes and delivering the programming via a virtual platform. The health coach will provide the Healthier Families modules either to individual child-parent pairs.
  Interventions: Behavioral: Healthier Families, COVID Edition; Behavioral: Teaching Kitchen Outreach

INTERVENTIONS:
Behavioral: Healthier Families, COVID Edition — Families randomized to this arm with receive12-weekly health coaching calls virtually with their family with topics such as nutrition, physical activity, sleep, and media use.
  Arms: Healthier Families, COVID Edition
Behavioral: Teaching Kitchen Outreach — Families receiving this intervention will recipe 11-weekly video recipes and groceries delivered to their door.

SUMMARY:
A randomized controlled trial enrolling 123 parent-infant dyads (English or Spanish speaking) comparing a virtual video Teaching Kitchen Outreach Program (TKO) with weekly grocery delivery (comparator group), to Healthier Families, COVID Edition (intervention group) which includes TKO plus a 12-week virtual health coaching intervention aimed at supporting family goal setting and behavior change including topics such as nutrition and physical activity.

DETAILED DESCRIPTION:
The aim of this work is to conduct a randomized controlled trial to test the effect of two evidenced based programs (Healthier Families and Teaching Kitchen Outreach (TKO) adapted to a virtual platform on improving family health.

Both the intervention and comparator condition receive up to 12 weekly short (about 2-3 minutes) Teaching Kitchen Outreach (TKO) videos. Recipe specific groceries are delivered to participants' homes by a third party grocery delivery company, and are available for pickup at a central location(s). These recipes reflect foods that can be purchased with SNAP and WIC and include tested meals and snacks that were developed and evaluated in person in Parks and Recreation after-school programming (Heerman W, Elsakary Y, Sommer E, Escarfuller J, Barkin S. Assessing the Scale and Spread of an Experiential Teaching Kitchen in After-School Programming Among School-Aged Children) through the long-standing Nashville Collaborative partnership (https://pediatrics.vumc.org/nashville-collaborative). Over more than a decade, the Nashville Collaborative has developed and tested programs together to improve health and wellness and reduce childhood obesity in the local community.

Those randomized to the intervention condition receive a 12-weekly health coach via a virtual platform (such as Zoom, FaceTime, or What's App) to provide an adapted version of the previously tested Healthier Families program. Adaptations include: shortening each session to 30 minutes and delivering the programming via a virtual platform. The health coach provides the Healthier Families modules to individual child-parent pairs. Any use of Zoom for participant participation will use a version of Zoom procured through Vanderbilt. The virtual version of Healthier Families was adapted from prior research in the Growing Right Onto Wellness (GROW) trial that worked with over 600 parent-child dyads and demonstrated a statistically significant effect on health behavior change (Barkin SL, Heerman WJ, Sommer EC, Martin NC, Buchowski MS, Schlundt D, Po'e EK, Burgess LE, Escarfuller J, Pratt C, Truesdale KP, Stevens J. Effect of a Behavioral Intervention for Underserved Preschool-Age Children on Change in Body Mass Index: A Randomized Clinical Trial).

ELIGIBILITY:
Inclusion Criteria:

* Currently participating in programming with one of the involved community partners, including, Parks and Recreation, Nashville Public Library, Project Transformation, Head Start, Martha O'Bryan, and St. Luke's; Patients who receive primary care at the Vanderbilt Primary Care Pediatrics Clinic are eligible as well.
* Parent/legal guardian age ≥ 18 years
* Parent legal guardian of a child ages 2-8
* Ability to participate on a virtual platform (such as Zoom, FaceTime, What's App, Google Hangouts)
* Ability to addend a Zoom tool training and complete a baseline survey prior to programming
* Be able to access virtual programming through online platforms, including YouTube
* Speak English or Spanish

Exclusion Criteria:

* Inability to complete data collection measures via telephone, Redcap, or paper measures
* Language other than English or Spanish

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 123 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2021-11-11 (Actual)

PRIMARY OUTCOMES:
Family Healthy Lifestyle Subscale | Baseline to 12 weeks
  The 6-item Family Healthy Lifestyle Subscale is a validated measure with higher scores indicating better family health (Crandall A, Weiss-Laxer NS, Broadbent E, et al. The Family Health Scale: Reliability and Validity of a Short- and Long-Form. Front Public Health. 2020;8:587125. doi:10.3389/fpubh.2020.587125). The total score ranges from 6-30 and is calculated by summing the responses to all 6 items of the Family Healthy Lifestyle Subscale. Each item uses a 5-point Likert scale ranging from 1 = "Strongly disagree" to 5 = "Strongly agree."

SECONDARY OUTCOMES:
Family Resilience and Connection Index | Baseline to 12 weeks
  The 6-item Family Resilience and Connection Index is a validated measure with higher scores indicating better family resilience and connection (Bethell CD, Gombojav N, Whitaker RC. Family Resilience And Connection Promote Flourishing Among US Children, Even Amid Adversity. Health Affairs (Millwood). 2019;38(5):729-737). doi:10.1377/hlthaff.2018.05425). The total Family Resilience and Connection Index score is calculated by summing the sub scores of 3 categories (score range in parentheses): Family resilience index (0-4), parent-child connection (0-1), and parent coping (0-1). For the family resilience index, 1 point was assigned for each time a parent responded "all of the time" to one of the 4 items. 1 point was assigned for each time a parent responded "very well" to the 2 items on parent-child connection and parent coping. The total score of the FRCI ranges from 0-6.

OTHER OUTCOMES:
Parent Nutrition Scale | Baseline to 12 weeks
  Parent nutrition was measured using the Starting the Conversation: Dietary Scale (Paxton AE, Strycker LA, Toobert DJ, Ammerman AS, Glasgow RE. Starting the conversation performance of a brief dietary assessment and intervention tool for health professionals. Am J Prev Med. 2011;40(1):67-71). It is a validated, 8-item instrument to assess diet, with lower scores indicating better nutrition. The total score ranges from 0-16.
Child Nutrition Food Categories | Baseline to 12 weeks
  Child nutrition was assessed based on participating children's 30-day consumption of six food categories from the CDC Dietary Screener, which contains items used widely on the Behavioral Risk Factor Surveillance System. Frequency of consumption within the following six food categories was analyzed: sugary beverages (combined soda and sweetened drinks), snacks, sweets, fruits, leafy greens, and other vegetables. The minimum score for each of the six defined food category was 0. There was no maximum score limit.
USDA Household Food Security Scale | Baseline to 12 weeks
  Food security was measured using a short form of the USDA Household Food Security Scale, which is a validated, 6-item instrument that categorizes households as food secure or food insecure (Blumberg SJ, Bialostosky K, Hamilton WL, Briefel RR. The effectiveness of a short form of the Household Food Security Scale. Am J Public Health. 1999;89(8):1231-4.). The total USDA Household Food Security score is calculated by summing the number of affirmative responses to each item. The total score ranges from 0-6. A total score less than 2 indicated no food insecurity or hunger. A total score of ≥ 2 indicated food insecurity. A total score of ≥ 5 indicated hunger.

CONTACTS AND LOCATIONS:
Overall Officials: Shari Barkin, MD, MSHS, Principal Investigator — Vanderbilt Univeristy Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Popescu F, Sommer EC, Mahoney MR, Adams LE, Barkin SL. Effect of a Virtual Home-Based Behavioral Intervention on Family Health and Resilience During the COVID-19 Pandemic: A Randomized Clinical Trial. JAMA Netw Open. 2022 Dec 1;5(12):e2247691. doi: 10.1001/jamanetworkopen.2022.47691. PMID 36538328